CLINICAL TRIAL: NCT07141394
Title: Coordinated Access for Addiction Recovery and Equity in VA Supportive Housing (CARE-VASH) (QUE 25-013)
Brief Title: Coordinated Access for Addiction Recovery and Equity in VA Supportive Housing
Acronym: CARE-VASH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QUX 25-001; QUE 25-013 (Other Grant/Funding Number: QUERI)
Record Dates: First submitted 2025-08-06; First posted 2025-08-26 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Homelessness; Substance Use Disorder (SUD)
Keywords: Homeless; Substance Use Disorder; Permanent Supportive Housing; Implementation Science
MeSH Terms: conditions — Substance-Related Disorders | interventions — Dosage Forms; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Investigators are implementing two evidence-based Substance Use Disorder (SUD) services - Medications for addiction treatment (MAT) and cognitive behavioral therapy for SUDs (CBT-SUD) - among Veterans in the Department of Housing and Urban Development-VA Supportive Housing Program (HUD-VASH).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Replicating Effective Programs (REP) (Experimental): A stakeholder-informed training and technical assistance implementation strategy
  Interventions: Drug: Medication for Addiction Treatment (MAT); Behavioral: Cognitive Behavioral Therapy for Substance Use Disorders (CBT-SUD)
- REP + Consumer Engagement (CE) (Active Comparator): REP plus CE package (educational materials, peer coaching, toolkit) to support MAT and CBT-SUD implementation.
  Interventions: Drug: Medication for Addiction Treatment (MAT); Behavioral: Cognitive Behavioral Therapy for Substance Use Disorders (CBT-SUD)
- Control Group (No Intervention): No MAT or CBT-SUD implementation

INTERVENTIONS:
Drug: Medication for Addiction Treatment (MAT) — MAT includes medications for alcohol use disorder (MAUD) and medications for opioid use disorder (MAUD). It reduces substance use, increases SUD treatment engagement, enhances quality of life, and reduces overdoses.
  Other Names: MAT
  Arms: REP + Consumer Engagement (CE); Replicating Effective Programs (REP)
Behavioral: Cognitive Behavioral Therapy for Substance Use Disorders (CBT-SUD) — An evidence-based psychotherapy that uses cognitive behavioral therapy to further recovery goals across SUD diagnoses.
  Other Names: CBT-SUD
  Arms: REP + Consumer Engagement (CE); Replicating Effective Programs (REP)

SUMMARY:
The Department of Housing and Urban Development-VA Supportive Housing (HUD-VASH) Program provides subsidized permanent housing with case management to homeless-experienced Veterans (HEVs). Up to 40% of Veterans exit HUD-VASH within two years of attaining housing; substance use disorders (SUDs) are one of the largest causes of returns to homelessness for HEVs. CARE-VASH QUERI proposes to implement and evaluate two evidence-based SUD services - Medications for addiction treatment (MAT) and cognitive behavioral therapy for SUDs (CBT-SUD) - among Veterans in HUD-VASH.

DETAILED DESCRIPTION:
The Department of Housing and Urban Development-VA Supportive Housing (HUD-VASH) program provides subsidized, permanent housing and supports to Veterans experiencing homelessness. Substance use disorders (SUDs) are a common primary or contributing factor to negative exits from HUD-VASH. The Coordinated Access for Addiction Recovery and Equity in VA Supportive Housing (CARE-VASH) QUERI will implement two evidence-based practices (EBPs) for SUDs-Medications for Addiction Treatment (MAT) and cognitive behavioral therapy for SUDs (CBT-SUD)-in 12 HUD-VASH sites. We will use the Replicating Effective Programs (REP) implementation bundle to support EBP implementation at all 12 sites. Half the sites (n=6) will also receive 9 months of consumer engagement (REP+CE). In a type 3 hybrid trial, we will use mixed methods to examine the impacts of REP vs. REP+CE. Using our trial data, we will develop a budget impact analysis and implementation playbook for our program partners to spread and sustain MAT and CBT-SUD in HUD-VASH.

ELIGIBILITY:
Inclusion Criteria:

* Homeless-experienced Veterans (HEVs) enrolled in the Department of Housing and Urban Development-VA Supportive Housing (HUD-VASH) Program.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7908 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach of MAT (Medications for Addiction Treatment) | 18 months post-implementation
  * (percent of) Veterans who used Medications for Opioid Use Disorder (MOUD) for OUD, ≥1 prescription
  * (percent of) Veterans who used MOUD for OUD for 180 days since initial prescription (without a break ≥14 days in supply)
  * (percent of) Veterans who used Medications for Alcohol Use Disorder (MAUD) for AUD, ≥1 prescription
  * (percent of) Veterans who used MAUD for AUD for 180 days since initial prescription (without a break ≥14 days in supply)
Reach of CBT-SUD (Cognitive Behavioral Therapy-Substance Use Disorders) | 18 months post-implementation
  * (percent of) Veterans with stimulant use disorder who had ≥1 visit for Cognitive Behavioral Therapy-Substance Use Disorders (CBT-SUD) or contingency management
  * (percent of) Veterans with substance use disorder with ≥1 CBT-SUD visit
  * (percent of) Veterans with substance use disorder with ≥9 CBT-SUD visits
Adoption of MAT (Medications for Addiction Treatment) | 18 months post-implementation
  % (percent of) Department of Housing and Urban Development - VA Supportive Housing (HUD-VASH) and mental health prescribers engaged with Veterans who ordered Medications for Opioid Use Disorder (MOUD) / Medications for Alcohol Use Disorder (MAUD) at least once
Adoption of CBT-SUD (Cognitive Behavioral Therapy-Substance Use Disorders) | 18 months post-implementation
  % (percent of) Department of Housing and Urban Development - VA Supportive Housing (HUD-VASH) case managers who delivered ≥1 CBT-SUD (Cognitive Behavioral Therapy-Substance Use Disorders) session
Sustainment of MAT (Medications for Addiction Treatment) | 18-27 months post-implementation
  * (percent of) Veterans who used Medications for Opioid Use Disorder (MOUD) for OUD, ≥1 prescription
  * (percent of) Veterans who used MOUD for OUD for 180 days since initial prescription (without a break ≥14 days in supply)
  * (percent of) Veterans who used Medications for Alcohol Use Disorder (MAUD) for AUD, ≥1 prescription
  * (percent of) Veterans who used MAUD for AUD for 180 days since initial prescription (without a break ≥14 days in supply)
  * (percent of) Department of Housing and Urban Development - VA Supportive Housing (HUD-VASH) and mental health prescribers engaged with Veterans who ordered Medications for Opioid Use Disorder (MOUD) / Medications for Alcohol Use Disorder (MAUD) at least once
Sustainment of CBT-SUD (Cognitive Behavioral Therapy-Substance Use Disorders) | 18-27 months post-implementation
  * (percent of) Veterans with stimulant use disorder who had ≥1 visit for Cognitive Behavioral Therapy-Substance Use Disorders (CBT-SUD) or contingency management
  * (percent of) Veterans with substance use disorder with ≥1 CBT-SUD visit
  * (percent of) Veterans with substance use disorder with ≥9 CBT-SUD visits
  * (percent of) Department of Housing and Urban Development - VA Supportive Housing (HUD-VASH) case managers who delivered ≥1 CBT-SUD (Cognitive Behavioral Therapy-Substance Use Disorders) session

SECONDARY OUTCOMES:
Housing retention | 1 year after implementation by cohort
  Difference in the mean days homeless over 1 year of follow-up for Veterans enrolled in trial sites that received the base versus enhanced implementation strategy, versus the expected number of days homeless had they enrolled in a comparison group of all sites not engaged in the trial
Provider experience | Baseline and 18 months post-implementation
  Experiences of and satisfaction with providing HUD-VASH services to HEVs with SUDs pre- and post- implementation, which will be assessed using semi-structured qualitative interviews (data will be coded from key findings in the narratives provided during the interviews).
Cost impact of Medications for Addiction Treatment (MAT) and Cognitive Behavioral Therapy-Substance Use Disorders (CBT-SUD) | 18 months (during the course of implementation)
  The predominant cost of delivering MAT in the Department of Housing and Urban Development-VA Supportive Housing (HUD-VASH) programs is prescriber time; for CBT-SUD, the predominant cost is case manager time. We will use VA administrative data to identify visits in which MAT was prescribed or CBT-SUD was delivered. Interviews with HUD-VASH prescribers will be used to estimate minutes/visit spent on MAT, including visits in which MAT was discussed but not prescribed; at implementation sites, we will add a mandated field to templated CBT-SUD notes that indicates time spent outside the encounter (e.g., preparing for the visit).
Acute care utilization | 1 year after implementation by cohort
  Emergency department visits and hospitalizations associated with primary SUD diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Emi Gabrielian, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Evelyn T Chang, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA; Erin P Finley, PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Emily Treichler, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol